CLINICAL TRIAL: NCT00914342
Title: A Cross-sectional Study on the Prevalence and Impact in Work Productivity of GERD in Primary Care Patients With Upper GI Symptoms Using the Novel Questionnaire GERD-Q. The Greek GERD-Q Study
Brief Title: Prevalence and Impact in Work Productivity of Gastroesophageal Reflux Disease (GERD) in Primary Care Patients With Upper Gastrointestinal (GI) Symptoms Using GerdQ
Acronym: GerdQ-Greece
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: AstraZeneca, AstraZeneca
Other Study IDs: NIS-GGR-DUM-2009/1
Record Dates: First submitted 2009-06-03; First posted 2009-06-05 (Estimated); Last update posted 2009-12-29 (Estimated); Status verified 2009-12

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: Gerd; GerdQ questionnaire; work productivity; Greece
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Upper-GI symptoms in primary-care patients

SUMMARY:
The purpose of the study is to provide data on the GERD prevalence as percentage of patients with upper GI symptoms that are identified with GERD using the GerdQ Questionnaire. Furthermore the study aims to estimate GERD prevalence in patients based on their symptoms as they respond to a physician's questionnaire, to observe possible variations between the two methods (physicians' symptom rating and GerdQ), to objectively measure treatment response and to identify the percentage of patients that may require alterations of their treatment. Finally, to describe the impact of GERD symptoms on work productivity.

ELIGIBILITY:
Inclusion Criteria:

* Patients with upper-GI symptoms the last week prior visiting the investigator

Exclusion Criteria:

* History of oesophageal, gastric or duodenal surgery
* Treatment with NSAIDs/Acetylsalicylic acid within the last week prior to the study visit
* PPI use for healing of NSAIDs induced ulcer or for HP eradication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who consult their primary care physician and have experienced upper-GI symptoms during the last week prior their consultation
Sampling Method: Probability Sample
Enrollment: 889 (Actual)
Dates: Start 2009-07; Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
GERD prevalence as percentage of patients with upper GI symptoms that are identified with GERD using the GerdQ Questionnaire (GerdQ score >=8). | Single Visit - once

SECONDARY OUTCOMES:
Estimation of GERD prevalence in patients based on their symptoms as they respond to a physician's questionnaire and to observe possible variations between the two methods (physicians' symptom rating and QerdQ) | Single Visit - Once
Describe the impact of GERD symptoms on work productivity. | Single Visit - Once
To objectively measure treatment response and to identify the percentage of patients that may require alterations of their treatment. | Single Visit - Once

CONTACTS AND LOCATIONS:
Overall Officials: Theodoros Rokkas, Dr, Principal Investigator — Henry Dynan Hospital, Athens, Greece; Panagiotis Pontikis, Dr, Study Director — AstraZeneca Greece
Locations (54):
- Greece (54):
  - Research Site, Pátrai, Achaias
  - Research Site, Mesologgion, Aitoloakarnaniaia
  - Research Site, Naupaktos, Aitoloakarnaniaia
  - Research Site, Grinion, Aitoloakarnania
  - Research Site, Aleksandroupoli, Aleksandroupoli
  - Research Site, Tripoli, Arkadias
  - Research Site, Acharnes, Attica
  - Research Site, Ag.Eleutherios, Attica
  - Research Site, Ag.Paraskeui, Attica
  - Research Site, Artémida, Attica
  - Research Site, Athens, Attica
  - Research Site, Chalandri, Attica
  - Research Site, Galatsi, Attica
  - Research Site, Glifada, Attica
  - Research Site, Ilipoli, Attica
  - Research Site, Kallithea, Attica
  - Research Site, Keratea, Attica
  - Research Site, Marousi, Attica
  - Research Site, N Makri, Attica
  - Research Site, N Smirni, Attica
  - Research Site, N.Herakeleios, Attica
  - Research Site, Peristeri, Attica
  - Research Site, Pikermi, Attica
  - Research Site, Pikerni, Attica
  - Research Site, Spata, Attica
  - Research Site, Chalcis, Chalkida
  - Research Site, Chalkidiki, Chalkidiki
  - Research Site, Chania, Chania
  - Research Site, Corinth, Corinth
  - Research Site, Mykonos, Cyclades
  - Research Site, Santorini, Cyclades
  - Research Site, Drama, Drama
  - Research Site, Zakynthos, Eptanisa
  - Research Site, Lamia, Ftiotida
  - Research Site, Heraklion, Herakleion
  - Research Site, Lexena, Ilias
  - Research Site, Véroia, Imathias
  - Research Site, Ioannina, Ioannina
  - Research Site, Karditsa, Karditsa
  - Research Site, Kastoria, Kastoria
  - Research Site, Katerini, Katerini
  - Research Site, Chrisoupoli, Kavala
  - Research Site, Komotini, Komotini
  - Research Site, Lakonia, Lakonia
  - Research Site, Larrisa, Larrisa
  - Research Site, Volos, Magnisia
  - Research Site, Kalamata, Mesinia
  - Research Site, Giannitsá, Pella
  - Research Site, Pereus, Pereus
  - Research Site, Ptolemaida, Ptolemaida
  - Research Site, Thessaloniki, Salonika
  - Research Site, Serres, Serres
  - Research Site, Trikala, Trikala
  - Research Site, Xánthi, Xanthi